CLINICAL TRIAL: NCT06213103
Title: Determining the Relevance of Mitochondrial Disease-associated ImmunoDeficiencies - MitoID
Brief Title: Mitochondrial Disease-associated ImmunoDeficiencies
Acronym: MitoID
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2022/36
Record Dates: First submitted 2023-06-09; First posted 2024-01-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Mitochondrial Disorders
Keywords: mitochondrial diseases; immunology; PBMCs; scATAC-seq; scRNA-seq
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- o Patient cohort: Patient with moleculary proven mitochondrial disorder
- o Control cohort: People without moleculary proven mitochondrial disorder

INTERVENTIONS:
Procedure: Patient cohort — Collection of 6 blood tubes at the inclusion visit.
Procedure: Control cohort — Collection of 6 blood tubes at the inclusion visit.

SUMMARY:
The study aims at characterizing the immune dysfunctions in patients with mitochondrial diseases. This has prognostic and diagnostic interest as well as potential for the discovery of new therapeutic strategies to alleviate disease burden.

DETAILED DESCRIPTION:
Mitochondrial pathologies are rare genetic diseases, and affect about 1 in 4300 people. These pathologies are characterized by an energetic deficit that can affect all organs, and can manifest from birth to adulthood. The clinical expression is very heterogeneous, the symptoms can include encephalopathies, myopathies, cardiomyopathies, among others, with frequently "an illegitimate association of symptoms" that add up in a progressive way. These pathologies are related to the presence of pathogenic mutations in the genes of the nuclear genome involved in mitochondrial metabolism, or directly in the genes of the mitochondrial DNA (mtDNA).

The immune system dysfunctions associated with mitochondrial diseases remain unknown to date despite the presence of the deleterious variant in leukocytes. Recent studies by group of the investigators and others in animal models clearly show the importance of mitochondrial functions in the regulation of inflammatory and antimicrobial processes. These experimental data are particularly relevant in light of recent clinical studies indicating that patients with mitochondriopathies have a higher rate of bacterial infections compared to control individuals.

The investigators hypothesized that immunological parameters assessment in patients will reveal new dysfunctions associated with these pathologies and that some of these parameters will be a prognostic factor in these "step-like" progression of these diseases.

This study will recruit 30 patients with mitochondrial disorders followed in Bordeaux University Hospital and Toulouse University Hospital for who the mutation of mitochondrial DNA has been previously identified. Among classical disease activity information, blood samples will be collected to study immunological parameters. Translational research will be realized on patient' samples to assess immune cell subsets and innate immune cells functions.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

  * Patient weighing more than 30kg
  * Person affiliated with or receiving a social security plan;
* Patient-specific inclusion criteria:

  * Patient with molecularly proven primary mitochondrial disease
  * Free, informed, written consent signed by parental authority holders for minor patients and the investigator prior to any examination required by the research and oral and/or written assent by the participant (depending on age).
  * Free, informed consent signed by the patient's representative for adult patients under guardianship and the investigator prior to any examination required by the research.
  * Free, informed consent signed by the patient of legal age and the investigator prior to any examination required by the research
* Specific inclusion criteria for controls:

  * Person who has been informed of the purpose of the study and person matched in age (+/- 5 years) and sex to a patient with primary mitochondrial disease at the time of sampling
  * Free, informed, and signed consent
  * Person with no known mitochondrial disease

Exclusion Criteria:

* Pregnant or breastfeeding women
* Refusal to consent to participate in research,
* Patients for whom molecular causes have not been formally identified (genetic analyses not performed, or no variant or variant of unknown significance after analysis).

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Patient cohort : Patient with moleculary proven mitochondrial disorder
  * Control cohort : People without moleculary proven mitochondrial disorder
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Immunological parameters | Inclusion visit
  Distribution of several quantitative immunological parameters at inclusion. The following parameters will be considered : Immunoglobulins in g/l (IgG subclasses, IgA, IgM)
Immunological parameters | Inclusion visit
  Distribution of several quantitative immunological parameters at inclusion. The following parameters will be considered : multiplex flow cytometry panels (Th1, Th2, Th17, Tfh, T, B, monocytes) in fluorescence intensity unit

SECONDARY OUTCOMES:
Immunological parameters | Inclusion visit
  Description of the percentage of patients with abnormal immunological parameters
infectious events | Inclusion visit
  Incidence of severe or recurrent infectious events retrospectively compared to the general population
Biological markers | Inclusion visit
  Description of the percentage of patients with abnormal key cytokines (TNF, IL-1b, IL-6, IL-12)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien TRIMOUILLE, MD, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - Chu Bordeaux, Bordeaux
  - Hopital Toulouse, Toulouse